CLINICAL TRIAL: NCT07126587
Title: Healthy Living Anson
Brief Title: Healthy Living Anson Study
Acronym: HLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Westat (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 24-2854; OT2HL158287 (NIH)
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-08

CONDITIONS: Obesity (Disorder); Diabetes Type 2; Heart Disease; Hypertension; Cancer; High Cholesterol
Keywords: Healthy Living Anson; HLA study; nutrition; healthy eating; overweight (BMI ≥ 25)
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Heart Diseases; Hypertension; Neoplasms; Hypercholesterolemia; Overweight | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Randomized delayed intervention control study - 4 months participants receive either the FIM intervention (healthy frozen meals, produce box, and education by a community health advocate (CHA)) or a physical activity (PA) education and support via a CHA. At the end of the 4 months, the FIM group will receive maintenance and the PA component, and the PA group receives the FIM component and continue for another 4 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Education and Food Delivery, Then Physical Activity Comparator (Experimental): Participants first receive nutrition counseling from a Community Health Advocate (CHA) and 10 biweekly healthy prepared meals for the first four weeks. For the next four weeks, participants will reduce to 6 biweekly healthy prepared meals and 2 produce boxes. After a 6 week break at midpoint, participants will receive peer supported physical activity counseling by a Community Health Advocate (CHA) and a mHealth text messaging for 8 weeks.
  Interventions: Behavioral: Nutrition Education and Food Delivery; Behavioral: Physical Activity Comparator
- Physical Activity Comparator, Then Nutrition Education and Food Delivery (Experimental): Participants first receive peer supported physical activity counseling by a Community Health Advocate (CHA) and a mHealth text messaging for 8 weeks. After a 6 week break at midpoint, participants will receive nutrition counseling by a Community Health Advocate (CHA) and 10 biweekly healthy prepared meals for the first four weeks. For the next four weeks, participants will reduce to 6 biweekly healthy prepared meals and 2 produce boxes.
  Interventions: Behavioral: Nutrition Education and Food Delivery; Behavioral: Physical Activity Comparator

INTERVENTIONS:
Behavioral: Nutrition Education and Food Delivery — Healthy frozen meals, produce boxes, and nutrition counseling
Behavioral: Physical Activity Comparator — Physical activity counseling, mHealth text messaging

SUMMARY:
The goal of this randomized delayed control intervention research study is to see if participants who receive education and healthy prepared meals improve the quality of their diet compared to participants who receive only physical activity education and coaching.

DETAILED DESCRIPTION:
Purpose: Evaluate whether a Food is Medicine (FIM) intervention improves the quality of food intake among rural adults who have at least one chronic disease or are at risk for chronic disease compared to those receiving a physical activity intervention.

Participants: English speaking Anson County residents 18 years or older

Procedures: Randomized delayed intervention control study design - 4 months receive either the FIM intervention (healthy frozen meals and/or produce box, and education by a Community Health Advocate (CHA) or physical activity (PA) education and support via a CHA. At the end of the 4 months, the FIM group will receive the PA intervention, and the PA group receives the FIM intervention with both groups continuing for another 4 months. Data collected will include a funder required survey (demographics, social, and behavioral factors) plus additional study related questions and biometrics. The survey will be completed online or in person for those requiring internet access or support. The biometrics will be obtained at an in-person session. Once enrollment is complete, participants will be randomized into either the FIM or PA group and receive their study materials. Data collection will occur at baseline, midpoint, and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants must be a resident of Anson County.
* At least 18 years of age.
* Have or be at risk for a chronic disease.
* Ability to make own dietary decisions.
* Ability to travel to a central Anson County location for data collection and group class sessions.
* Ability and willingness to try the prepared meals.
* Ability to store 10 frozen meals in a freezer.
* Ability to communicate in English
* No dietary restrictions or food allergies such that a Mediterranean diet is not appropriate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Med-South Dietary Risk Assessment Score | Baseline, Midpoint (Month 4), Endpoint (up to Month 10)
  The Med-South Dietary Risk Assessment (DRA) is scored as the sum of the column score for each numbered item, with column score multiplied by 0.5 for Items 3.3 and 3.4. The score ranges from 0 to 10, 0 meaning no adherence and 10 meaning full adherence. With regard to diet quality, the first response option is considered "desirable," the second "could be improved," and the third "needs to be improved.

SECONDARY OUTCOMES:
Physical Activity Questionnaire | Baseline, Midpoint (Month 4), Endpoint (Up to Month 10)
  Assessed by the International Physical Activity Questionnaire (IPAQ) - Short Form. This questionnaire is a well-validated 7-day physical activity recall assessment for physical activity. This will measure frequency (days per week) and duration (time per day) for each specific type of activity. Three specific activity types will be scored, walking, moderate-intensity activity, and vigorous-intensity activity. Participants will be scored based on metabolic equivalent of task units (MET, energy expenditure). This will be determined by multiplying the frequency by duration (in hours). Each activity type will have MET calculated separately, and the summation of each score will generate the the overall physical activity score in MET units. Scores will range from 0-99. We will only report the overall score. Higher scores indicate higher levels of physical activity and more energy expenditure.
Skin Carotenoids | Baseline, Midpoint (month 4), Endpoint (up to month 10)
  Description: Skin carotenoid level is a number from 0 to 800 that approximates carotenoids in the skin. A Veggie Meter uses reflection spectroscopy to determine the level of skin carotenoids using the fingertip. Measurements are taken three times, with scores being averaged and reported. A higher score indicates more fruit and vegetable intake.
Nutrition Insecurity | baseline, endpoint
  Nutrition Insecurity will be measured using a survey with one item. This item indicates the frequency in which a participant has skipped or cut the size of meals due to lack of finances. Frequency is established using a likert scale, always to never, with one selection option. Always would signify high nutrition insecurity, and never would signify low nutrition insecurity.

CONTACTS AND LOCATIONS:
Overall Officials: Anissa I Vines, MS, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.